CLINICAL TRIAL: NCT01581307
Title: A Phase II Clinical Trial Evaluating Overall Survival With Therasphere® In Conjunction With 2nd-Line FOLFOX In Patients With Gemcitabine-Refractory Pancreatic Carcinoma With Liver Metastases
Brief Title: Phase II Trial Evaluating OS With Therasphere® + 2nd-Line FOLFOX in Pancreatic Liver Mets
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: BTG International Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-16764
Record Dates: First submitted 2012-04-18; First posted 2012-04-20 (Estimated); Results first posted 2017-01-06 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2016-11

CONDITIONS: Liver Cancer; Pancreatic Cancer
Keywords: liver; pancreas; chemotherapy; radiotherapy
MeSH Terms: conditions — Liver Neoplasms; Pancreatic Neoplasms | interventions — Leucovorin; Fluorouracil; Oxaliplatin; Folfox protocol; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2nd Line Chemotherapy With Radiotherapy (Experimental): Administration of 2nd line chemotherapy will consist of a modified FOLFOX7 (Folinic acid, 5-Fluorouracil, and Oxaliplatin) will take place at least 2 weeks after the completion of first-line chemotherapy. Generally, second-line chemotherapy is given every two weeks for 6-10 cycles.
  The goal of treatment with TheraSpheres is to allow a large dose of radiation to be delivered directly to the tumor(s) with less risk of toxic effects from radiation to other parts of the body or to healthy liver tissue.
  Interventions: Drug: FOLFOX7 (Folinic acid, 5-Fluorouracil, and Oxaliplatin); Device: TheraSpheres

INTERVENTIONS:
Drug: FOLFOX7 (Folinic acid, 5-Fluorouracil, and Oxaliplatin) — The usual treatment if gemcitabine chemotherapy has failed is chemotherapy with a drug combination called FOLFOX (folinic acid, 5-FU and oxaliplatin) given through a vein every 2 weeks for 6-10 cycles. Participants will receive this treatment.
  Other Names: Leucovorin; LV; FOL; OX; 5-Fluorouracil (5-FU); FOLFOX; ELOXATIN
Device: TheraSpheres — TheraSpheres are a medical device containing yttrium-90 (Y-90), a radioactive material that has been used previously in the treatment of liver tumors. Y-90 is incorporated into very tiny glass beads called microspheres and is injected into the liver through the blood vessels supplying the liver. TheraSpheres have restricted approval from the United States Food and Drug Administration (FDA) for the treatment of hepatocellular liver cancer; but has not yet been approved for the treatment of pancreatic cancer that has spread to the liver.
  Other Names: radiotherapy; radioembolization

SUMMARY:
The purpose of this study is to evaluate the safety and impact on survival with treatment with 90-Y glass microspheres in conjunction with leucovorin, 5-fluorouracil (5-FU) and oxaliplatin (FOLFOX) as second-line treatment with in patients gemcitabine-refractory metastatic pancreatic cancer with predominantly liver metastases.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have metastatic pancreatic cancer with predominantly liver metastatic disease (> 50%), as determined by the principal investigator (PI0 and referring medical oncologist that have progressed on gemcitabine-based chemotherapy.
* Patients can have solitary, multifocal unilobar, or bilobar disease.
* Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 2
* No prior radiation or embolization of the liver
* Childs-Pugh score ≤ 7
* Lung shunting that predicts lung dose to be ≤ 30 Gy in a single treatment
* The effects of TheraSpheres on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because radioactive spheres are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document
* Adequate baseline hematopoietic function:

  * total white blood cell count equal to or greater than 3,000/mm^3
  * absolute granulocyte count greater than 1,500/mm^3
  * platelet count equal to or greater than 50,000/mm^3
  * Hemoglobin > 8.0

Exclusion Criteria:

* Patients currently receiving any other investigational agents
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because TheraSpheres are radioactive and radiation is a known agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with TheraSpheres, breastfeeding should be discontinued if the mother is treated with TheraSpheres.
* Initiation of second-line chemotherapy not consisting of FOLFOX
* Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy. In addition, antiretrovirals are known radiation sensitizers and could dramatically increase the risk of fulminant hepatic failure. Therefore, human immunodeficiency virus(HIV)-positive patients are excluded from the study because of possible lethal side effects.
* Bulk disease (tumor volume > 70% of the target liver volume)
* Aspartic transaminase (AST) or alanine transaminase (ALT) > 5 times upper limit of normal (ULN)
* Bilirubin > 2 mg/dL
* Child-Pugh score > 7
* Tumor volume > 50% of liver combined with an albumin < 3 g/dL
* Complete occlusion of main portal vein causing portal hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-04; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Hoffe, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at Moffitt Cancer Center June 2012 through March 2014.
Groups:
- 2nd Line Chemotherapy With Radiotherapy: Administration of 2nd line chemotherapy will consist of a modified FOLFOX7 (Folinic acid, 5-Fluorouracil, and Oxaliplatin) will take place at least 2 weeks after the completion of first-line chemotherapy. Generally, second-line chemotherapy is given every two weeks for 6-10 cycles.
  The goal of treatment with TheraSpheres is to allow a large dose of radiation to be delivered directly to the tumor(s) with less risk of toxic effects from radiation to other parts of the body or to healthy liver tissue.
  FOLFOX7 (Folinic acid, 5-Fluorouracil, and Oxaliplatin): The usual treatment if gemcitabine chemotherapy has failed is chemotherapy with a drug combination called FOLFOX (folinic acid, 5-FU and oxaliplatin) given through a vein every 2 weeks for 6-10 cycles. Participants will receive this treatment.
  TheraSpheres: TheraSpheres are a medical device containing yttrium-90 (Y-90), a radioactive material that has been used previously in the treatment of liver tumors.
Period: Overall Study
Arm/Group | 2nd Line Chemotherapy With Radiotherapy
Started | 9
Completed | 8
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All participants. Outcome Measures may reference participants evaluable at time of analysis.
Groups:
- 2nd Line Chemotherapy With Radiotherapy: Administration of 2nd line chemotherapy consisted of a modified FOLFOX7 (Folinic acid, 5-Fluorouracil, and Oxaliplatin) to take place at least 2 weeks after the completion of first-line chemotherapy. Generally, second-line chemotherapy was to be given every two weeks for 6-10 cycles.
Arm/Group | 2nd Line Chemotherapy With Radiotherapy
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 5
Age, Continuous [Median (Full Range); unit: years] | 70.44 [57 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Median Overall Survival (OS)
Description: OS, defined as the time from study enrollment to death from any cause, will be analyzed and summarized with the survival probabilities over time using Kaplan-Meier method. Confidence intervals for the median OS rates at different time points will be constructed when appropriate.
Time Frame: Up to 29 months
Population: All participants evaluable at time of analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 2nd Line Chemotherapy With Radiotherapy
Number analyzed (Participants) | 8
months | 14.09 [1.379 to 27.79]

2. Secondary Outcome: Rate of Progression Free Survival (PFS)
Description: PFS defined as the time from study enrollment to progression in the liver by modified Response Evaluation Criteria in Solid Tumors (RECIST) or death, whichever occurs first will be analyzed and summarized with the survival probabilities over time using Kaplan-Meier method. Confidence intervals for the median PFS rates at different time points will be constructed when appropriate.
Time Frame: Up to 29 months
Population: All participants evaluable at time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | 2nd Line Chemotherapy With Radiotherapy
Number analyzed (Participants) | 8
Participants | 3

3. Secondary Outcome: Overall Response Rate (ORR)
Description: The overall response: ORR = complete response (CR) + partial response (PR). Rate will be summarized using both point estimates and exact confidence intervals based on the binomial distribution by groups.
Time Frame: Up to 29 months
Population: All participants evaluable at time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | 2nd Line Chemotherapy With Radiotherapy
Number analyzed (Participants) | 7
Participants
  Complete Response | 0
  Partial Response | 5

ADVERSE EVENTS:
Time Frame: 30 months
Description: All Adverse Events (AEs) and Serious Adverse Events (SAEs) are reported regardless of causality.
Arm/Group | 2nd Line Chemotherapy With Radiotherapy
Serious Adverse Events (participants affected / at risk) | 5/9
Other Adverse Events (participants affected / at risk) | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2nd Line Chemotherapy With Radiotherapy (N=9)
Anemia (Blood and lymphatic system disorders) | 3 (5)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (6)
Bloating (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (3)
Gastric hemorrhage (Gastrointestinal disorders) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify - melena (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3)
Death NOS (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Fever (General disorders) | 2 (3)
Malaise (General disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Biliary tract infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (2)
Blood bilirubin increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 2 (3)
White blood cell decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2)
Confusion (Psychiatric disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hot flashes (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2nd Line Chemotherapy With Radiotherapy (N=9)
Anemia (Blood and lymphatic system disorders) | 4 (14)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (3)
Watering eyes (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (14)
Bloating (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 4 (5)
Flatulence (Gastrointestinal disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify - stool color changes (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (6)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Mucositis oral (Gastrointestinal disorders) | 3 (5)
Dry mouth (Gastrointestinal disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 4 (4)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (10)
Chills (General disorders) | 2 (2)
Fever (General disorders) | 2 (2)
Malaise (General disorders) | 1 (1)
General disorders and administration site conditions - Other, thrush (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Hepatobiliary disorders - Other, jaundice (Hepatobiliary disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Biliary tract infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Lymphocyte count decreased (Investigations) | 8 (36)
Alkaline phosphatase increased (Investigations) | 6 (7)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Alanine aminotransferase increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 2 (2)
INR increased (Investigations) | 2 (2)
Weight loss (Investigations) | 2 (3)
Weight gain (Investigations) | 1 (3)
Blood bilirubin increased (Investigations) | 3 (6)
Neutrophil count decreased (Investigations) | 7 (13)
Platelet count decreased (Investigations) | 6 (17)
White blood cell decreased (Investigations) | 7 (23)
Investigations - Other, Prothrombin time increased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 4 (7)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (15)
Hyponatremia (Metabolism and nutrition disorders) | 5 (18)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (9)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (23)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal and connective tissue disorders - Other, muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 4 (5)
Headache (Nervous system disorders) | 4 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4)
Dysgeusia (Nervous system disorders) | 2 (2)
Memory impairment (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2)
Skin and subcutaneous tissue disorders - Other, discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)
Hypertension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes